CLINICAL TRIAL: NCT02237222
Title: Evaluation of the Gait Performance Measures 'Functional Mobility Scale' and 'Gillette Functional Assessment Questionnaire' in Children With Neuromuscular Diagnoses
Brief Title: Evaluation of Gait Performance in Children With Neuromuscular Diagnoses
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: GaitPerformance_2014
Record Dates: First submitted 2014-09-01; First posted 2014-09-11 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Psychometrics of Two Translated Measurement Tools
Keywords: Outcome Assessment; Gait; Neuromuscular Diseases; Psychometrics; Clinical Assessment Tools
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gait rehabilitation: Multi-modal therapy program including physiotherapy with the aim of gait improvement, Lokomat or treadmill training, strength training, sports therapy.
  Frequency and intensity are individually assigned.
  Interventions: Other: Gait rehabilitation

INTERVENTIONS:
Other: Gait rehabilitation

SUMMARY:
The aims of this project are to evaluate the psychometric properties of the German versions of the two performance questionnaires 'Functional Mobility Scale' (FMS) and 'Gillette Functional Assessment Questionnaire - walking scale' (GFAQ) in children between 6-18 years with a neuromuscular diagnosis.

DETAILED DESCRIPTION:
The German versions of the two questionnaires 'Functional Mobility Scale' (FMS) and 'Gillette Functional Assessment Questionnaire - walking scale' (GFAQ) are evaluated in terms of construct validity, inter- and intra-rater reliability as well as responsiveness in children with a neuromuscular diagnosis, who absolve an inpatient stay in the rehabilitation center of the University Chilren's Hospital Zurich, Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Neuromuscular diagnosis
* Age: 6-18 years
* Rehabilitation goal = improvement of walking abilities

Exclusion Criteria:

* Children's whose parents are not German-speaking

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with neuromuscular diagnoses, who are inpatients in the rehabilitation center of the University Children's Hospital Zurich in Affoltern am Albis.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Functional Mobility Scale (FMS) | Participants will be followed for the duration of the rehabilitation stay, an expected average of 12 weeks, with measurements at admission and discharge.
  The questionnaire is filled in independently by the parents, the primary nurse as well as the physiotherapist of each child.
Gillette Functional Assessment Questionnaire - Walking Scale (GFAQ) | Participants will be followed for the duration of the rehabilitation stay, an expected average of 12 weeks, with measurements at admission and discharge.
  The questionnaire is filled in independently by the parents, the primary nurse as well as the physiotherapist of each child.

SECONDARY OUTCOMES:
Global Rating Scale (GRS) | Participants will be followed for the duration of the rehabilitation stay, an expected average of 12 weeks, with only one measurement at discharge.
  A global rating on the perceived change of the child's functional mobility over the rehabilitation period and whether this change is perceived as meaningful or not; on a 5-point Likert scale, scored by the parents and the physiotherapist.

OTHER OUTCOMES:
Functional Independence Measure for Children (WeeFIM) | Participants will be followed for the duration of the rehabilitation stay, an expected average of 12 weeks, with measurements at admission and discharge.
  The WeeFIM-Item Locomotion (Walking) is scored by the primary nurse.
10-Meter Walk Test (10MWT) | Participants will be followed for the duration of the rehabilitation stay, an expected average of 12 weeks, with only one measurement at discharge.
  For the evaluation of the construct validity of the FMS and the GFAQ, the 10MWT comfortable speed as well as maximal speed will be performed shortly before discharge on a 14-meter long track with standardized instructions.
6-Minute walk test (6MinWT) | Participants will be followed for the duration of the rehabilitation stay, an expected average of 12 weeks, with only one measurement at discharge.
  For the evaluation of the construct validity of the FMS and the GFAQ, the 6MinWT is performed shortly before discharge on a 30-meter long track with standardized instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Ammann-Reiffer, MPTSc, Principal Investigator — University Children's Hospital Zurich, Rehabilitation Center Affoltern
Locations (1):
- University Children's Hospital Zurich, Rehabilitation Center, Affoltern am Albis, Switzerland